CLINICAL TRIAL: NCT04294849
Title: Exercise Intolerance and Skeletal Muscle Bioenergetics in Children With Deep Venous Thrombosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study enrollment ceased because this was enrolling as a pilot study until a larger study (FUVID) was submitted, approved and received funding.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ayesha Zia, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU-2019-1406
Record Dates: First submitted 2020-02-13; First posted 2020-03-04 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Magnetic Resonance Spectroscopy; Exercise Test; Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venous Thromboembolism Arm (Experimental): This will be a cohort of patients age 8- ≤ 21 years old with objectively diagnosed DVT and/or PE.
  Interventions: Other: Magnetic Resonance Imaging; Other: Bicycle Ergometry; Other: Lab Panel; Behavioral: Questionnaires

INTERVENTIONS:
Other: Magnetic Resonance Imaging — A. Phosphorous 31 MR Spectroscopy to evaluate skeletal muscle metabolism via measurement of depletion and recovery of phosphocreatine (PCr) B. Non-invasive arterial spin labeling MRI to evaluate lymphatic flow velocities and venous flow
Other: Bicycle Ergometry — To measure peak VO2 as a representation of global aerobic fitness
Other: Lab Panel — A. Inflammatory lab panel (IL-6, IL-8, TNF alpha, P-selectin, high sensitivity CRP, IL-6 receptor, TNF R1/R2) drawn at diagnosis B. Thrombin Generation Assay to measure hypercoagulability and Thromboelastography prior to initiating anticoagulation
Behavioral: Questionnaires — A. Dalhousie Dyspnea Scale B. Godin Leisure Time Exercise Questionnaire C. Pediatric Venous Quality of Life Questionnaire

SUMMARY:
This is a prospective cohort study of 30 patients who are 8-21 years of age with venous thromboembolism (VTE)- either lower extremity deep venous thrombosis (DVT) or pulmonary embolism (PE).

DETAILED DESCRIPTION:
Participants will be in three groups- those with lower extremity DVT, those with PE, or those with both lower extremity DVT and PE. Patients will have blood drawn for thrombin generation assay, thromboelastography assay, and thromboinflammatory panel in addition to standard of care labs for diagnosis of VTE and management of anticoagulation. The patients will then fill out questionnaires on quality of life and level of exercise at their first outpatient visit 4 weeks after diagnosis. At approximately 3-6 months after diagnosis, patients will undergo two days of testing for the research study. All patients will have exercise testing using bicycle ergometry to measure global aerobic fitness. They will once again fill out questionnaires about their quality of life and level of physical activity. After a 24 hour rest period, DVT patients will undergo 31P-MR Spectroscopy and non-invasive spin labeling MRI to provide data on skeletal muscle bioenergetics (phosphocreatine metabolism), and lymphatic and venous flow respectively in the affected leg compared to the unaffected leg. This will allow each patient to be his or her own control. After these research procedures, patients will continue to receive standard of care treatment for their VTE in the Bleeding and Thrombosis clinic.

ELIGIBILITY:
Inclusion Criteria:

* Age 8- ≤ 21 years old AND
* Lower extremity deep venous thrombosis OR
* Lower extremity deep venous thrombosis AND pulmonary embolism OR
* Pulmonary Embolism

Exclusion Criteria:

* Contraindications to exercise, such as post-surgical patients with cast immobility or fractures
* Patients unable to follow instructions/commands at baseline due to developmental delay
* Patients with congenital heart disease and abnormal pulmonary circulation/perfusion
* Contraindications to undergoing magnetic resonance imaging

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Phosphocreatine Depletion and Recovery | 31P MR Spectroscopy will be performed one time between 3-6 months after diagnosis.
  Phosphocreatine (PCr) will be measured at baseline, during performance of submaximal exercise to fatigue and then at rest in the 31 P MR Spectroscopy Scan.
Assessment for Venous Occlusion | Arterial Spin labeling MRI will be performed one time between 3-6 months after diagnosis.
  Arterial spin labeling MRI will be utilized to examine venous flow in bilateral lower extremities to assess for venous occlusion.
Assessment of Lymphatic flow | Arterial Spin labeling MRI will be performed one time between 3-6 months after diagnosis
  Arterial spin labeling MRI will be utilized to assess lymphatic flow in bilateral lower extremities to assess for adequate lymphatic drainage.
Inflammatory markers | Diagnosis to 4 weeks.
  A custom blood assay will be used to assess inflammation at the time of the thrombotic event. Assay will include measurements of IL-6, IL-8, TNF-alpha, CRP, IL-10, IL-6 receptor, TNF alpha receptors.
Coagulation markers | Diagnosis to 4 weeks.
  Thrombin generation assay (TGA) will be used to assess hypercoagulability, and thromboelastography will be used to assess fibrinolysis. These will be drawn at the time of the thrombotic event.

SECONDARY OUTCOMES:
Exercise Intolerance | Pulmonary embolism patients will undergo this testing at 4-6 weeks after diagnosis. Deep venous thrombosis only patients will undergo testing at 3 months.
  Participants will undergo Cardiopulmonary Exercise testing to assess maximal aerobic fitness.
Godin Leisure Time Activity Questionnaire | Questionnaire to be filled out to assess activity at baseline, then one month after diagnosis, and 3-6 months after diagnosis.
  Patients will be asked to fill out a questionnaire to determine levels of physical activity for comparison at different time points throughout treatment.
Pediatric Venous Quality of Life Questionnaire | Participants will be asked to fill this questionnaires 4 weeks after diagnosis, and 3-6 months after diagnosis.
  Questionnaire to determine quality of life in various areas including school, leisure time, home, and relationships with peers.
OSA-18 Sleep Apnea Questionnaire | Participants will be asked to fill out this questionnaire at one month post diagnosis.
  Patients will be asked to complete this questionnaire to assess sleep quality and screen for obstructive sleep apnea.
PHQ-9 Questionnaire | Participants will be asked to fill this questionnaire one month after diagnosis.
  Participants will fill out this questionnaire to screen for depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Zia, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center / Children's Medical Center, Dallas, Texas, United States